CLINICAL TRIAL: NCT01300000
Title: Effects of Early Nutrient Intake on Growth and Body Composition
Brief Title: Effects of Early Nutrition on Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Collaborators: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK65
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Infant Newborn
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Human Milk (Active Comparator): ad lib
  Interventions: Other: Human Milk
- Milk based standard infant formula (Active Comparator): ad lib
  Interventions: Other: Milk based standard infant formula
- Milk based investigational infant formula (Experimental): ad lib
  Interventions: Other: Investigational infant formula

INTERVENTIONS:
Other: Human Milk — ad lib
  Arms: Human Milk
Other: Investigational infant formula — ad lib
  Arms: Milk based investigational infant formula
Other: Milk based standard infant formula — ad lib
  Arms: Milk based standard infant formula

SUMMARY:
The primary objective of the study is to compare the growth of infants fed standard infant formula with infants fed a reduced calorie and protein formula.

ELIGIBILITY:
Inclusion Criteria:

* good health
* singleton birth with gestational age 37-42 weeks
* infant's birth weight >or = to 2500 grams
* exclusive breastfeeding or exclusively formula feeding
* within a defined geographical boundary
* mother has no problems communicating in English

Exclusion Criteria:

* adverse maternal, fetal or infant medical history
* congenital disease or malformation affecting growth or development
* illness or social problems in mother or infant
* temporary residents

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 649 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Weight gain | 1- 365 days

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 1-365 days
Infant Anthropometrics | 1 - 365 days; 24 months

OTHER OUTCOMES:
Vascular | at 24 months
Maternal Anthropometrics | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Marriage, PhD, Study Chair — Abbott Nutrition
Locations (1):
- MRC Childhood Nutrition Research Center, Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831